CLINICAL TRIAL: NCT04924946
Title: Current Use in Intensive Care Units by Intensivists of Antihypertensive Drugs
Acronym: CUICUI-AHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191137
Record Dates: First submitted 2021-04-29; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-04

CONDITIONS: Antihypertensive Drugs in ICU
Keywords: intensive care; antihypertensive drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs — * Time to monitor blood pressure values in target targets
  * Need for administration of another antihypertensive drug
  * Disappearance of organ failure attributable to hypertension
  * Weaning from an extra-renal purification
  * Weaning from mechanical ventilation
  * Improved kidney function
  * Iatrogenic hypotension
  * Need for suspension of treatment
  * Other side effect

SUMMARY:
Multicenter, prospective and observational study of practices and impacts of the use of antihypertensive therapies in intensive medicine and intensive care

DETAILED DESCRIPTION:
Multicenter, prospective observational cohort study on 200 patients, by doctor's questionnaire on the prescription of antihypertensive drugs in intensive care, follow-up over 72 hours of the prescription.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Admitted to an intensive care unit
* Patient having presented a state of circulatory shock, defined by the need for continuous administration of a vasopressive amine for at least one hour, among: Noradrenaline, Adrenaline
* In whom the introduction of drug treatment for antihypertensive purposes is decided

Exclusion Criteria:

* Patient admitted to intensive care for a hypertensive emergency (hypertensive surge or malignant arterial hypertension leading to organ dysfunction
* Patient who has already received at least one anti-hypertensive drug during his stay in intensive care
* Cerebro-injured patient, proven or suspected cerebral edema, head trauma <1 month, decrease in cerebral perfusion measured
* Proven or suspected active bleeding
* Patient refusal of participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients hospitalized in intensive care
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Make an inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs in intensive care and intensive care settings | 60 days after inclusion
  Description in number of drugs
Make an inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs in intensive care and intensive care settings | 60 days after inclusion
  Description in percentage of drugs
Make an inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs in intensive care and intensive care settings | 60 days after inclusion
  therapeutic classes
Make an inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs in intensive care and intensive care settings | 60 days after inclusion
  administration methods
Make an inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs in intensive care and intensive care settings | 60 days after inclusion
  prescription chronology
Make an inventory of prescribing habits and detect any differences in efficacy and tolerance of antihypertensive drugs in intensive care and intensive care settings | 60 days after inclusion
  reasons for prescribers

SECONDARY OUTCOMES:
Search for efficiency differences between the different molecules | 60 days after inclusion
  Time to control blood pressure values in the targeted targets
Search for efficiency differences between the different molecules | 60 days after inclusion
  Need for administration of another antihypertensive drug
Search for efficiency differences between the different molecules | 60 days after inclusion
  Disappearance of organ failure attributable to hypertension
Search for efficiency differences between the different molecules | 60 days after inclusion
  Weaning from an extra-renal purification
Search for efficiency differences between the different molecules | 60 days after inclusion
  Weaning from mechanical ventilation
Search for efficiency differences between the different molecules | 60 days after inclusion
  Improved kidney function
Search for differences in side effects between the different molecules | 60 days after inclusion
  Iatrogenic hypotension
Search for differences in side effects between the different molecules | 60 days after inclusion
  Need for suspension of treatment
Search for differences in side effects between the different molecules | 60 days after inclusion
  Other side effect

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Intensive Care Victor Dupouy Hospital, Argenteuil
  - Intensive Care Avicenne Hsopital, Bobigny
  - Intensive Care Louis Mourier Hospital, Colombes
  - Intensive Care Longjumeau Hospital, Longjumeau
  - Intensive Care Bichat Hospital, Paris
  - Intensive Care René Dubos Hospital, Pontoise
  - Intensive Care Tours Hospital, Tours

IPD SHARING:
Plan to Share IPD: No